CLINICAL TRIAL: NCT06872970
Title: Outcomes of Open Reduction and Internal Fixation of Femoral Neck Fractures Using Dynamic Hip Screw Vs Cannulated Screws and Medial Buttress Plate
Brief Title: Open Reduction in Femoral Neck Fractures
Acronym: OR FNFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samer youssef mansour meglaa (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Samer youssef mansour meglaa, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Open reduction
Record Dates: First submitted 2025-02-16; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-04

CONDITIONS: Femoral Neck Fractures
Keywords: Open reduction
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: Using watson-jones or smith-peterson approach in open reduction of femoral neck fractures then fixation of fractures by dynamic hip screws vs cannulated screws and medial butteess plate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open reduction of femoral neck fractures in healthy adults (Experimental): Open reduction of femoral neck fractures in healthy adults between 16 years and 60 years old using cannulated screws and medial buttress plate through watson jones or smith peterson approach
  Interventions: Procedure: Open reduction of femoral neck fractures and internal fixation by dynamic hip screws; Procedure: Open reduction of femoral neck fractures using watson jones or smith peterson approachand internal fixation by cannulated screws and medial buttress plate
- Open reduction of femoral neck fractures (Experimental): Open reduction and internal fixation of femoral neck fracture in healthy adults between 16 years and 60 years old using dynamic hip screw through watson jones or smith peterson approach
  Interventions: Procedure: Open reduction of femoral neck fractures and internal fixation by dynamic hip screws; Procedure: Open reduction of femoral neck fractures using watson jones or smith peterson approachand internal fixation by cannulated screws and medial buttress plate

INTERVENTIONS:
Procedure: Open reduction of femoral neck fractures and internal fixation by dynamic hip screws — Open reduction of femoral neck using watson jones or smith peterson approach fractures then fixation of fractures by dynamic hip screws
Procedure: Open reduction of femoral neck fractures using watson jones or smith peterson approachand internal fixation by cannulated screws and medial buttress plate — Open reduction of femoral neck fractures then fixation of fractures by cannulated screws and medial buttress plate

SUMMARY:
Outcomes of open reduction and internal fixation of femoral neck fractures using dynamic hip screw versus cannulated screws combined with medial buttress plate.

DETAILED DESCRIPTION:
-Femoral neck fractures (FNFs) in patients under the age of 50 years account for less than 5% of all hip fractures and are typically the result of a high-energy event.

FNFs in young patients, particularly displaced fractures, are challenging to treat. Internal fixation remains the consensus, and the quality of the reduction is more important than the time to surgery.

Femoral head necrosis and fracture nonunion have always been the two major complications of femoral neck fracture treatment, which greatly increases the difficulty of treatment and places a high burden on social and medical resources.

As previous studies have demonstrated, reoperation rate for a failure of internal fixation ranges from 10% to 48.8% and has remained largely unchanged over the past 30 years.

There are many options to treat femoral neck fracture. Previous studies reported that femoral neck fractures with following surgery are associated implant failure.

Currently, the most common types of fixation include cannulated screws, hip screw systems, proximal femur plates, and cephalomedullary nails. [7]

Arthroplasty may be an option for elderly patients, but is generally not feasible for young patients; young patients with FNF require a more durable and promising fixation. However, there is no consensus on the best fixation method for FNF in young patients.

CS has better biomedical properties such as anti-rotation and less invasive, which was widely used in non-displaced intracapsular fractures.

DHS could maintain the neck-shaft angle and anatomical reduction, which is helpful for fracture fixation.

A medial buttress plate can clamp the fracture apex, neutralize shearing forces, and transfer them into compressive forces into the plane of cannulated screws or other typical construct.

Thus far, there has been no optimal internal fixation method.

ELIGIBILITY:
Inclusion Criteria:

* patients of both genders between the ages of 16 to 60 years old and had trauma caused femoral neck fracture.
* patients of both genders with Garden's type three and four femoral neck fractures

Exclusion Criteria:

* patients of both genders below the age of 16 and above 60 years old.
* patients with pathological femoral neck fractures.
* patients with autoimmune diseases like rheumatoid arthritis.
* patients with neglected femoral neck fractures(more than 1 week).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Harris hip score | 3 years
  Using harris hip score evaluate to evaluate post operative:
  1. pain
  2. amount and type of support
  3. limp
  4. distance walked
  5. shoes and socks
  6. sitting
  7. climbing stairs

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Keshet D, Bernstein M. Open Reduction Internal Fixation of Femoral Neck Fracture-Anterior Approach. J Orthop Trauma. 2020 Aug;34 Suppl 2:S27-S28. doi: 10.1097/BOT.0000000000001818. PMID 32639347